CLINICAL TRIAL: NCT07105527
Title: Dexmedetomidine During Carotid Endarterectomy: a Registry on Safety and Satisfaction of Patients and Operators (DexTEA)
Status: Completed | Type: Observational
Sponsor: Saint Camillus International University of Health Sciences (Other)
Responsible Party: Principal Investigator, Diego Fiume, Principal Investigator, Saint Camillus International University of Health Sciences
Other Study IDs: 0002376
Record Dates: First submitted 2025-07-11; First posted 2025-08-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hypertension Arterial; Desaturation; Bradycardia; Surgery (Major Vascular); Hypotension During Surgery; Dexmedetomidine Induced Sedation; Fentanyl Analgesia; Satisfaction, Patient; Satisfaction, Personal; Nausea/Vomiting
Keywords: dexmedetomidine; cervical plexus block; sedation; satisfaction; humans; follow-up; prospective study; endarterectomy; clamping time; analgesic
MeSH Terms: conditions — Hypertension; Bradycardia; Patient Satisfaction; Personal Satisfaction; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sedation with 1 mcg/kg fentanyl + 0.03 mg/kg midazolam in boluses: until RASS -1/-2
- sedation with dexmedetomidine 1 mcg/kg/h for 10 minutes and then 0.3-0.5 mcg/kg/h: until RASS -1/-2

SUMMARY:
From an anesthesiological perspective, carotid endarterectomy (CEA) is an operation that is increasingly being performed with locoregional techniques and sedation. The aim of this observational study was to compare dexmedetomidine with midazolam and fentanyl during CEA in terms of perioperative adverse events, patient, anesthetist, and surgeon satisfaction, as well as the possible reduction in clamping time and the number of times additional local anaesthesia is needed.

Sixty patients listed for CEA were enrolled and two types of sedation were used, both protocols widely used in our hospital, resulting in the formation of two groups of patients. Both the intermediate and superficial cervical plexus blocks were administered, and the patients in Group 1 were sedated with midazolam and fentanyl, and Group 2 was sedated with dexmedetomidine. The investigators examined comorbidities, surgical time and clamping, and possible intraoperative use of local anaesthetics and intraprocedural complications, and follow-up at 180 days to observe any residual deficits. The data were analysed with Statistical Package for Social Science (SPSS) Statistics 25 (IBM).

DETAILED DESCRIPTION:
Carotid endarterectomy (CEA) is one of the most common procedures in vascular surgery, along with lower limb revascularization, and endovascular surgery. It has long been considered a standard for the treatment of carotid artery disease; it is currently considered the most valid medical approach for significantly decreasing the risk of ischemic stroke in symptomatic patients and a 'quasi standard' for the treatment in patients with high-grade carotid stenosis. From an anesthesiological perspective, it is a procedure than can be approached in different ways, i.e., with the patient under a state of general anaesthesia or with locoregional techniques (with possible sedation).

Although the recent General Anesthesia vs. Local Anesthesia (GALA) trial did not demonstrate the superiority of either of the above mentioned anaesthesiological management methods for this type of surgery, there are differences between the two techniques, including the risk of postoperative cognitive impairment.

Considering the type of surgery, for greater control of haemodynamic management without excessive hypotension or hypertension, at our Unit (Sant'Eugenio Hospital, Rome, Italy), the surgery is performed through the locoregional approach, sedating the patient only to keep it still during the procedure but awake to be able to evaluate haemodynamic compensation.

Under locoregional anaesthesia, a standard for anesthesia in this procedure is the intermediate cervical| plexus block. The cervical plexus block provides anaesthesia and analgesia for neck and head surgery, including CEA procedures. Usually, along with peripheral blockade, the use of hypnotics with a sedative dosage is preferred to increase patient compliance. There are numerous drugs used to sedate patients during a procedure, starting with the most widely used drugs, such as midazolam and propofol, followed by the most recently introduced drug, dexmedetomidine. The latter is a well-known superselective a2-agonist drug with hypnotic, sedative, anxiolytic, sympatholytic and analgesic activity that suppresses the neuronal noradrenergic cascade at the locus coeruleus level without inducing respiratory depression. It has no rebound effects even after 24 hours of continuous infusion and, therefore, lends itself well to administration even for short-term procedures. It also possesses a good safety margin. The purpose of this observational study is to compare the two major sedation techniques and protocols currently used and the usefulness of dexmedetomidine during carotid endarterectomy in terms of minor and major adverse events and patient, anaesthetist, and surgeon satisfaction, as well as the possible reduction in clamping time and the number of times the surgeon needs to administer additional local anaesthesia.

Study Design and Population A single-center, prospective observational study was conducted entirely within the Sant'Eugenio Hospital. All methods were performed in accordance with the guidelines and regulations of the Declaration of Helsinki, and this prospective observational study was approved by the Independent Ethics Committee of the Sant'Eugenio Hospital. Written informed consent was obtained from all patients whose data were collected. The minimum target set to start the study was the enrolment of 60 patients to be divided equally into two groups, since our group of anesthetists uses, without preference, two sedation protocols, in addition to cervical plexus blockade, for TEA operations in vascular surgery, both of which are approved in the literature and in internal hospital procedures. This process took place from January 2021 to December 2023. All patients referred to the Vascular Surgery of the hospital who were candidates for carotid endoarterectomy surgery were considered eligible for the study. The exclusion criteria included: severe liver failure (Child-Pugh classes B or C) or severe hypoproteinemia (albuminemia < 3.0 g/di); age <18 yr; baseline heart rate <50 bpm; Il or Ill grade atrioventricular block without a pacemaker; malignant hyperthermia suspected or established; psychiatric disorders; emergency surgery, inability to provide consent for tie procedure.

Endpoints The study has primary endpoints and secondary endpoints. Primary endpoints: An anaesthetist and surgeon evaluated the usefulness of dexmedetomidine during carotid endarterectomy in terms of minor and major adverse events and patients, anaesthetists and surgeons' satisfaction. This evaluation was carried out on a graded scale from 1 to 4 (4=very satisfied, 3=satisfied, 2=slightly satisfied, 1=not satisfied), which was specifically used for this observational study.

The secondary endpoints were possible reduction in clamping time and the number of times the surgeon had to administer local anaesthesia (in our study, 0.5% lidocaine).

Anaesthesia protocol In the preprocedural phase, after signing the informed consent, the patient was cannulated with peripheral venous access and a peripheral artery for monitoring. In accordance with the perioperative fluid management in the Enhanced Recovery After Surgery (ERAS) protocol, the patient fasted with clear fluid for at least two hours before induction of anaesthesia, and Ringer's lactate was used to maintain volemia.

All patients were given a nerve block of both the intermediate and superficial cervical plexus with an ultrasound-guided needle using levobupivacaine 0.33% + mepivacaine 1.5% as a local anaesthetic, for a total volume of 15ml. The block was executed when the patient was fully awake and collaborating; in case of excessive agitation, a premedication with Midazolam 0,03 mg/kg for a maximum of 2 mg was used.

Once the preliminary phase was completed, the investigators took note of the type of sedation chosen between the two methods under analysis that are both used in our hospital, the choice of sedation protocol was at the discretion of the attending anesthetist. To standardize the procedure, for drug dosages, in addition to in-house protocols, data from the literature were used.

* GROUP 1: standard sedation with 1 mcg/kg fentanyl + 0.03 mg/kg midazolam in boluses until a Richmond Agitation-Sedation Scale (RASS) equivalent to -1/-2 was achieved.
* GROUP 2: sedation with dexmedetomidine 1 mcg/kg/h for 10 minutes and then 0.3-0.5 mcg/kg/h until RASS -1/-2.

Sedation was initiated once vital parameters were stabilized on the operating table, until the end of surgical procedure.

Typically, once on the operating table, the patient was started on continuous monitoring of cardiac, respiratory and neurological activity. At the end of surgery, the patient was then monitored over the following 4 hours in the recovery room and discharged according to Aldrete's criteria, noting the discharge times for each patient.

Data collection The data were collected from individual patient records. These included physical status, medical history, American Society of Anesthesiologists (ASA) risk score assessment, home therapy, any adverse events recorded during previous anaesthesia, recent blood test results, recent EKG and preoperative imaging (chest X-ray), if necessary. For this study, the following data were examined: medical history of comorbidities present, surgical time, clamping time, percentage of shunts and conversion to general anaesthesia, any intraoperative use of local anaesthetics (lidocaine 0.5 %), intraprocedural complications and follow-up at 180 days to observe any residual deficits.

Statistical analysis To assess the best sample size, the investigators calculated it on the number of patients with carotid pathology referred to the vascular surgery department, with a 95% confidence interval and a 5% margin of error. The study involved the enrolment of 60 patients, divided into two groups according to the anaesthesia performed in the operating room, who were compared according to the parameters assessed and recorded.

Statistical analysis was performed using chi-square tests and Fisher's exact tests for comparing proportions and Student's t tests for comparing means ÷ Standard Deviation (SD). A P value <0.05 was considered to indicate statistical significance. Statistical analysis was performed using IBM SPSS Statistics 25 (IBM).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were candidates for carotid endoarterectomy elective surgery
* Age >18yr
* Ability to provide consent for the procedure

Exclusion Criteria:

* severe liver failure (Child-Pugh classes B or C) or severe hypoproteinemia (albuminemia < 3.0 g/dl)
* age <18yr
* baseline heart rate <50 bpm; II or III grade atrioventricular block without a pacemaker
* malignant hyperthermia suspected or established
* psychiatric disorders
* emergency surgery
* inability to provide consent for the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The minimum target set to start the study was the enrolment of 60 patients to be divided equally into two groups, since our group of anaesthetists uses, without preference, two sedation protocols, in addition to cervical plexus blockade, for TEA operations in vascular surgery, both of which are approved in the literature and in internal hospital procedures
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Patients, anaesthetists and surgeons' satisfaction | Periprocedural
  evaluation on a graded scale from 1 to 4 (4=very satisfied, 3=satisfied, 2=slightly satisfied, 1=not satisfied),
Number of Participants with Hypertension | Periprocedural
  Systolic Blood Pressure> 145 mmHg
Number of Participants with Hypotension | Periprocedural
  Systolic Blood Pressure <100 mmHg
Number of Participants with Bradycardia | Periprocedural
  Heart Rate <50 beats per minute
Number of Participants with Nausea and/or Vomiting | Periprocedural
  Number of events
Number of Participants with Desaturation | Periprocedural
  Hemoglobin saturation <88%
Number of Participants with Chronic surgical site pain | Up to 6 months
  Numerical Rating Scale (NRS): Zero is equivalent to no pain and 10 indicates the worst possible pain

SECONDARY OUTCOMES:
Change in clamping time | Periprocedural
  time (minutes)
Number of times the surgeon had to administer local anaesthesia | Periprocedural
  number of times the surgeon had to administer local anaesthesia (in our study, 0.5% lidocaine)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Fiume, MD PhD, Study Chair — UniCamillus - Saint Camillus International University of Health and Medical Sciences
Locations (1):
- Sant'Eugenio Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD); however, anonymized data may be made available upon reasonable request, subject to sponsor approval and ethical considerations.

REFERENCES:
- [Background] Malek LA, Malek AK, Leszczynski J, Toutounchi S, Elwertowski M, Spiewak M, Domagala P. Carotid clamping time as a risk factor for early restenosis after carotid endarterectomy. Eur J Vasc Endovasc Surg. 2005 Aug;30(2):143-6. doi: 10.1016/j.ejvs.2005.04.023. PMID 15936960
- [Background] Do W, Cho AR, Kim EJ, Kim HJ, Kim E, Lee HJ. Ultrasound-guided superficial cervical plexus block under dexmedetomidine sedation versus general anesthesia for carotid endarterectomy: a retrospective pilot study. Yeungnam Univ J Med. 2018 Jun;35(1):45-53. doi: 10.12701/yujm.2018.35.1.45. Epub 2018 Jun 30. PMID 31620570
- [Background] McCutcheon CA, Orme RM, Scott DA, Davies MJ, McGlade DP. A comparison of dexmedetomidine versus conventional therapy for sedation and hemodynamic control during carotid endarterectomy performed under regional anesthesia. Anesth Analg. 2006 Mar;102(3):668-75. doi: 10.1213/01.ane.0000197777.62397.d5. PMID 16492813
- [Background] Bekker AY, Basile J, Gold M, Riles T, Adelman M, Cuff G, Mathew JP, Goldberg JD. Dexmedetomidine for awake carotid endarterectomy: efficacy, hemodynamic profile, and side effects. J Neurosurg Anesthesiol. 2004 Apr;16(2):126-35. doi: 10.1097/00008506-200404000-00004. PMID 15021281
- [Background] Sidorowicz M, Owczuk R, Kwiecinska B, Wujtewicz MA, Wojciechowski J, Wujtewicz M. Dexmedetomidine sedation for carotid endarterectomy. Anestezjol Intens Ter. 2009 Apr-Jun;41(2):78-83. PMID 19697824
- [Background] Reel B, Maani CV. Dexmedetomidine. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK513303/ PMID 30020675
- [Background] Ramos-Matos CF, Bistas KG, Lopez-Ojeda W. Fentanyl. 2023 May 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459275/ PMID 29083586
- [Background] Dyck JB, Maze M, Haack C, Vuorilehto L, Shafer SL. The pharmacokinetics and hemodynamic effects of intravenous and intramuscular dexmedetomidine hydrochloride in adult human volunteers. Anesthesiology. 1993 May;78(5):813-20. doi: 10.1097/00000542-199305000-00002. PMID 8098190
- [Background] Rahimzadeh P, Faiz SHR, Imani F, Derakhshan P, Amniati S. Comparative addition of dexmedetomidine and fentanyl to intrathecal bupivacaine in orthopedic procedure in lower limbs. BMC Anesthesiol. 2018 Jun 6;18(1):62. doi: 10.1186/s12871-018-0531-7. PMID 29875020
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Nacif-Coelho C, Correa-Sales C, Chang LL, Maze M. Perturbation of ion channel conductance alters the hypnotic response to the alpha 2-adrenergic agonist dexmedetomidine in the locus coeruleus of the rat. Anesthesiology. 1994 Dec;81(6):1527-34. doi: 10.1097/00000542-199412000-00029. PMID 7992922
- [Background] Rossel T, Kersting S, Heller AR, Koch T. Combination of high-resolution ultrasound-guided perivascular regional anesthesia of the internal carotid artery and intermediate cervical plexus block for carotid surgery. Ultrasound Med Biol. 2013 Jun;39(6):981-6. doi: 10.1016/j.ultrasmedbio.2013.01.002. Epub 2013 Mar 15. PMID 23499343
- [Background] Ramachandran SK, Picton P, Shanks A, Dorje P, Pandit JJ. Comparison of intermediate vs subcutaneous cervical plexus block for carotid endarterectomy. Br J Anaesth. 2011 Aug;107(2):157-63. doi: 10.1093/bja/aer118. Epub 2011 May 24. PMID 21613278
- [Background] Perisanidis C, Saranteas T, Kostopanagiotou G. Ultrasound-guided combined intermediate and deep cervical plexus nerve block for regional anaesthesia in oral and maxillofacial surgery. Dentomaxillofac Radiol. 2013;42(2):29945724. doi: 10.1259/dmfr/29945724. Epub 2012 Aug 29. PMID 22933534
- [Background] Pandit JJ, Satya-Krishna R, Gration P. Superficial or deep cervical plexus block for carotid endarterectomy: a systematic review of complications. Br J Anaesth. 2007 Aug;99(2):159-69. doi: 10.1093/bja/aem160. Epub 2007 Jun 18. PMID 17576970
- [Background] Heyer EJ, Gold MI, Kirby EW, Zurica J, Mitchell E, Halazun HJ, Teverbaugh L, Sciacca RR, Solomon RA, Quest DO, Maldonado TS, Riles TS, Connolly ES Jr. A study of cognitive dysfunction in patients having carotid endarterectomy performed with regional anesthesia. Anesth Analg. 2008 Aug;107(2):636-42. doi: 10.1213/ane.0b013e3181770d84. PMID 18633045
- [Background] Zdrehus C. Anaesthesia for carotid endarterectomy - general or loco-regional? Rom J Anaesth Intensive Care. 2015 Apr;22(1):17-24. PMID 28913451
- [Background] Hynes N, Sultan S. Carotid Surgery Is the Gold Standard for High-Risk (HRP) Carotid Artery Intervention: Five-Year Cost-Effectiveness and Quality Stroke-Free Survival Comparison Between Carotid Endarterectomy (CEA), Carotid Angioplasty, and Stenting Technique (CAST), and Optimal Medical Therapy (OMT). J Vasc Surg. 2011 Feb;53(2):558
- [Background] GALA Trial Collaborative Group; Lewis SC, Warlow CP, Bodenham AR, Colam B, Rothwell PM, Torgerson D, Dellagrammaticas D, Horrocks M, Liapis C, Banning AP, Gough M, Gough MJ. General anaesthesia versus local anaesthesia for carotid surgery (GALA): a multicentre, randomised controlled trial. Lancet. 2008 Dec 20;372(9656):2132-42. doi: 10.1016/S0140-6736(08)61699-2. Epub 2008 Nov 27. PMID 19041130
- [Background] Ferguson GG, Eliasziw M, Barr HW, Clagett GP, Barnes RW, Wallace MC, Taylor DW, Haynes RB, Finan JW, Hachinski VC, Barnett HJ. The North American Symptomatic Carotid Endarterectomy Trial : surgical results in 1415 patients. Stroke. 1999 Sep;30(9):1751-8. doi: 10.1161/01.str.30.9.1751. PMID 10471419
- [Background] North American Symptomatic Carotid Endarterectomy Trial Collaborators; Barnett HJM, Taylor DW, Haynes RB, Sackett DL, Peerless SJ, Ferguson GG, Fox AJ, Rankin RN, Hachinski VC, Wiebers DO, Eliasziw M. Beneficial effect of carotid endarterectomy in symptomatic patients with high-grade carotid stenosis. N Engl J Med. 1991 Aug 15;325(7):445-53. doi: 10.1056/NEJM199108153250701. PMID 1852179

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT07105527/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT07105527/ICF_001.pdf